CLINICAL TRIAL: NCT02179684
Title: Surgery or Clinical Follow-up in Patients With Bell's Palsy. A Prospective, Parallell, Single Center, Randomized , Open Surgery Clinical Study.
Brief Title: Surgery or Clincial Follow up, in Patients With Bell' s Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Malou Hultcrantz, M.D. Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bell´sPalsy
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Bell Palsy
Keywords: Cranial Nerve fascial paresis
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early surgery (Experimental): Patienst with Bell´s Palsy with an early surgical intervention (< 3month), according to 'baby-sitter' method
  Interventions: Procedure: Baby-sitter surgery N. fascialis
- Conventional treatment and follow-up (Active Comparator): Patienst with Bell´s Palsy treated with conventional treatment and standardized physiotherapy according to Jaqueline Diels model.
  Interventions: Other: Conventional treatment and follow-up

INTERVENTIONS:
Procedure: Baby-sitter surgery N. fascialis
  Arms: Early surgery
Other: Conventional treatment and follow-up — Patient´s with Bells´palasy are treated with conventional treatment and follow-up
  Arms: Conventional treatment and follow-up

SUMMARY:
The purpose of this study is to investigate if an early surgical intervention on patienst with Bell´s Palsy has a better impact on their facial muscular function and their quality of life as compared to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Bell´s Palsy
2. Men and women aged 18-55 y
3. Score < 70 according to Sunny Brook scale (SB)
4. Signed informed consent

Exclusion Criteria:

1. High bloodpressure
2. Diabetes
3. Pregnancy
4. Currently on immunodepressive treatment
5. Smoker
6. Psychiatric disorder
7. Cor incomp, according to NYHA grade: IV, kidney or liver disorder, that greatly influence patienst ability to receive surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-02 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Sunny Brook (SB) score > 70 | 1 year
  Patients with Bell´s Palsy that has been randomized to conventional treatment or early surgical intervention are scored according to SB after 12 month of study participation.

SECONDARY OUTCOMES:
Facial Disability Index | 15 month
  Change in Facial Disability Index
FaCe | 15 month
  Change in FaCe quality score

CONTACTS AND LOCATIONS:
Overall Officials: Malou Hultcrantz, M.D prof., Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm, Solna
  - Uppsala Akademiska Hospital, EENT department, Uppsala, Uppsala County